CLINICAL TRIAL: NCT01394705
Title: FITT Exercise Counseling With Interactive Accelerometry and Physical Activity in Adolescents at Increased Risk of Early Cardiovascular Disease: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Tracy Curran, Clinical Exercise Physiologist, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P00000416
Record Dates: First submitted 2011-06-14; First posted 2011-07-14 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Coronary Artery Disease Risk High
Keywords: patients at increased risk for atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (No Intervention): standard of care (office provider exercise counseling)
- Intervention (Experimental): The intervention group received a personalized exercise prescription (using the FITT principles) and wore an accelerometer up to 7days/week (most waking hours) and logged their activity by regularly (3 times a week) uploading the device for a period of 3 months, use of the internet was supervised by a parent or guardian. Their activity was monitored via the online BodyMedia site on a regular basis by study personnel and feedback was provided at least once a week through email and/or phone calls
  Interventions: Device: BodyMedia

INTERVENTIONS:
Device: BodyMedia — Accelerometer
  Arms: Intervention

SUMMARY:
This pilot study seeks to compare the change in energy expenditure and fitness levels of patients seen in the Children's Hospital Preventive Cardiology program receiving standard of care provider exercise counseling to similar patients receiving Frequency, Intensity, Time, Type (FITT) exercise prescription and counseling combined with BodyMedia supported by an online interactive tool.

The investigators primary hypothesis is that this interactive technology coupled with support from a exercise specialist will increase the energy expenditure of the investigators patients over standard of care provider counseling.

The investigators Secondary hypotheses include greater improvement in measured physical fitness Peak oxygen consumption (VO2max), oxygen consumption (VO2) at anaerobic threshold (AT) and ventilation/carbon dioxide (VE/VCO2) slope, lipid profiles, blood pressure, arterial stiffness, body mass index (BMI), BMI percentile, and self-efficacy in the intervention group compared to control.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at increased risk of atherosclerosis based on lipid profiles (Total Cholesterol > 199 mg/dL, High Density Lipoprotein < 40 mg/dL, LDL > 129 mg/dL, blood pressure (Systolic Blood Pressure or Diastolic Blood Pressure > 90th percentile), obesity (>85%Body Mass Index)
2. Ages 13-21 years
3. Reporting an average of less than 60 minutes per day of moderate to vigorous exercise most (5) days of the week.
4. Regular access to the internet with the capacity to download the device
5. Commitment on the part of a parent to supervise internet access as part of this protocol

Exclusion Criteria:

1. Unable to exercise based on physician recommendations or medical conditions
2. Unable/unwilling to complete requirements of the research study including consent and assent.
3. Not proficient in English

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2011-06; Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy c Curran, MS, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Childrens Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 38 completed study, 21 randomized to each group, 2 lost to follow-up in each group with an N of 19 in each group.
Groups:
- Standard of Care; Intervention: BodyMedia: Accelerometer
Period: Overall Study
Arm/Group | Standard of Care | Intervention
Started | 21 | 21
Completed | 19 | 19
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Intervention | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 17 | 33
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 15.7 [13.1 to 20.3] | 15.9 [12.7 to 21.8] | 15.8 [12.7 to 21.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 15 | 16 | 31
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 14 | 19 | 33
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity
Description: Total time (minutes) in Physical Activity in one week
Time Frame: Baseline, 3 months
Measure: Median (Full Range); unit: minutes per week
Groups:
- Standard of Care: office provider exercise counseling
- Intervention: BodyMedia: Accelerometer wear
Arm/Group | Standard of Care | Intervention
Number analyzed (Participants) | 19 | 19
minutes per week
  Baseline | 457 [19 to 2343] | 443 [71 to 1219]
  Follow-up | 364 [0 to 2037] | 279 [0 to 1266]
Statistical Analysis 1: Comparison: Standard of Care vs Intervention; Test type: Superiority; p = .65, Fisher Exact
Statistical Analysis 2: Comparison: Standard of Care vs Intervention; Test type: Superiority; p = 0.65, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Body Mass Index
Description: Secondary hypotheses include greater improvement in body mass index (BMI) reported below.
Time Frame: Baseline, 3 months
Measure: Median (Full Range); unit: BMI (kg/m2)
Arm/Group | Standard of Care | Intervention
Number analyzed (Participants) | 19 | 19
BMI (kg/m2)
  Baseline | 30 [17 to 64] | 33 [19 to 49]
  Follow up | 30 [16 to 67] | 32 [19 to 50]
Statistical Analysis 1: Comparison: Standard of Care vs Intervention; Test type: Superiority; p = 0.76, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Study participant data was collected for 3 months.
Arm/Group | Standard of Care | Intervention
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-04-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT01394705/Prot_SAP_000.pdf